CLINICAL TRIAL: NCT05941663
Title: Microbiome Development in the Early Healing of Osseointegrated Implants. Impact of Surface Composition (SLActive® vs. SLA® Surface)
Brief Title: Microbiome Development in the Early Healing of Osseointegrated Implants
Acronym: PiMicrobiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: URI 104-210623
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Microbiota; Dental Implants

STUDY DESIGN:
Intervention Model Description: Split mouth design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The assessment and the measurements were performed by a separate person, not the operator. The patient did not know in which quadrant SLActive® or SLA® implants were placed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLAactive (Experimental): Implants provided were Bone Level Tapered (Bone Level Tapered) Roxolid® implants with a SLActive® surface
  Interventions: Other: Dental implant surface
- SLA (Active Comparator): Implants provided were Bone Level Tapered (Bone Level Tapered) Roxolid® implants with a SLA® surface
  Interventions: Other: Dental implant surface

INTERVENTIONS:
Other: Dental implant surface — Implants provided were Bone Level Tapered (Bone Level Tapered) Roxolid® implants with a SLActive® or SLActive® surface

SUMMARY:
The aim is to compare the microbiome composition on the first month of healing and 2 years after rehabilitation in two different implant surfaces (SLA® vs SLActive®). Subjects in need of two or more dental implants (canine to molars) in two different quadrants will be included so that, one study test (SLActive®) and one study control (SLA®) implant will be placed in different quadrants in healed extraction sites. Gingival crevicular fluid (GCF) samples will be taken for microbiome analysis at different time points. Samples will be processed using high throughput sequencing technologies (Illumina® MiSeq) and the raw sequencing reads will be processed with the Quantitative Insights Into Microbial Ecology (QIIME2) pipeline. DADA2 will be used for quality trimming and inferring amplicon sequence variants (ASVs). Taxonomy will be assigned to ASVs using the Naive Bayesian Classifier integrated in QIIME2 plugins and the eHOMD RefSeq database. Alpha-diversity and Beta diversity will be calculated and measured. Differences in bacterial abundance will be analyzed using linear models for differential abundance analysis (LinDA).

This is the long-term follow-up of the randomized clinical trial entitled "Randomized controlled study to evaluate the clinical behavior of dental implants with SLActive® surface vs. SLA® surface" Promoter Code: CR 2017-05, Internal Code: 18/580-R_P, Promoter: Institute Straumann AG. In this new protocol, the participants included in the clinical trial at the Complutense University of Madrid will be selected, who will undergo a new follow-up visit at 2 years, to measure the clinical, radiographic and microbiological situation. periodontal treatment without any additional intervention. In addition, it is intended to analyze the microbiome of the samples of gingival crevicular fluid that we have frozen from the patients of the UCM, as well as of the samples that are taken after two years. All these changes are promoted by our ETEP (Etiology and Therapeutics of Periodontal and Peri-implant Diseases) research group, independently of the original sponsor of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, at least 18 years old
* Partially edentulous patients rehabilitated with at least two dental implants (canine to molars) placed in two different quadrants in healed sites (3 months post extraction) as part of the previous RCT.
* Subject must have voluntarily signed the informed consent, are willing and able to attend scheduled follow-up visits, and agree that the encoded data will be collected and analyzed.

For the current investigation, only those participants treated in the University Complutense of Madrid (n=30) will be selected

Exclusion Criteria:

* Any contraindications for oral surgical procedures
* Dental implant placement contraindicated according to Instructions for Use (IFU)
* Subjects with inadequate oral hygiene (FMPS ≥ 20%)
* Subjects who are currently heavy smokers (defined >10 cigarettes per day or >1 cigar per day) or who use chewing tobacco
* Subjects with drug or alcohol abuse
* Patients requiring soft tissue and bone grafting procedures
* Patients having had soft tissue grafting procedures within the last 3 months and bone grafting procedures within the last 6 months in the region where a study implant is planned
* Keratinized soft tissue height of less than 2 mm where a study implant is planned
* Inadequate bone volume
* Severe bruxism or clenching habits
* Woman who are pregnant or planning to become pregnant at any point during the study duration.
* Patients who have systemic factors that could interfere with the healing process of either bone or soft tissue or the osseointegration process (e.g. bone metabolism disturbances, uncontrolled diabetes mellitus, anticoagulation drugs/ hemorrhagic diatheses)
* Patients with local factors that could interfere with the healing process, such as untreated periodontal diseases, acute infection of implant site, temporomandibular joint disorders, treatable pathologic diseases of the jaw and changes in the oral mucosa)
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.

Patients will be informed verbally and in written paper of the visit at 2-year post-implant placement, and will need to sign a new informed consent for this evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Microbiome composition | 2 years
  Samples will be processed by sequencing the 16S rRNA gene V3-V4 hypervariable region using MiSeq (Illumina, CA)

SECONDARY OUTCOMES:
Radiographic measurements | 2 years
  The reference point for the bone level measurement is the implant shoulder. The bone level will be measured as the distance between the implant shoulder and the first visible bone contact on the implant. The bone level will be measured on the mesial and distal aspect of the 2 study implants. Mean bone level changes between two time-points will be computed by subtracting the average bone level from one visit with the other.
Peri-implant diseases incidence | 2 years
  A full periodontal chart will be recorded of each patient at visit 10 (2 years after implant placement). Probing pocket depth, recession, bleeding on probing, plaque presence on 6 sites per tooth/implant will be registered (mesial, medial and distal, at buccal and lingual sides). This will be performed with a North Carolina Periodontal Probe and values will be given in millimeters
Questionnaire of oral care | 2 years
  A questionnaire about the maintenance and oral care that the patient has followed during the last 2 years will be recorded in order to better understand the information obtained from clinical, radiographical and microbiological parameters. The following questions will be asked: (1) Did you receive periodontal maintenance care in the last 6 months? (2) How many appointments for maintenance care have you accomplished in the last 2 years? (3) Do you use interproximal devices for your everyday oral care? (4) Did you received peri-implant or periodontal non-surgical therapy in the last 2 years? And surgical? This information will be completed by searching in the individual history of the data recording system of the university.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University Complutense of Madrid (UCM), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided